CLINICAL TRIAL: NCT06468566
Title: Identification of Benign and Malignant Breast Nodules Using Opalogram Ultrasonography: A Multicenter Study
Brief Title: Identification of Benign and Malignant Breast Nodules Using Ultrasound-modulated Optical Tomography: A Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Xin-Wu Cui (Other)
Collaborators: Hubei Cancer Hospital (Other); Guangxi National Hospital (Unknown); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor-Investigator, Xin-Wu Cui, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2024(S044)
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer Female
Keywords: Ultrasonic light scattering imaging; Breast Cancer; Metastasis; Artificial intelligence
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Whether to use ultrasound light scattering imaging equipment
  Interventions: Diagnostic Test: Ultrasound light scattering imaging equipment
- Conventional ultrasound
- Device Assistant physician
  Interventions: Diagnostic Test: Ultrasound light scattering imaging equipment

INTERVENTIONS:
Diagnostic Test: Ultrasound light scattering imaging equipment — Radiologists use ultrasound light scattering imaging to evaluate the benign and malignant nature of breast nodules
  Groups: Device Assistant physician; Whether to use ultrasound light scattering imaging equipment

SUMMARY:
Ultrasonic light scattering imaging is a new functional imaging technology that combines traditional B-mode ultrasound imaging and light scattering tomography (DOT). It can improve the accuracy of early diagnosis of breast cancer based on the characteristics of abnormal blood supply and oxygen consumption of lesions. This study aims to evaluate the value of ultrasonic light scattering imaging in the differential diagnosis of benign and malignant breast nodules, and to evaluate the consistency between ultrasonic light scattering imaging and examiners in the differential diagnosis of benign and malignant breast nodules.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women and the second leading cause of cancer death worldwide. Therefore, early detection and timely treatment of breast cancer are of great significance to controlling and reducing breast cancer mortality. Breast ultrasound has been widely used in the detection of breast cancer, but ultrasound is highly dependent on the examiner in terms of technology, and the examination results are greatly affected by the examiner's subjectivity, which increases unnecessary surgery and punctures, causing great trouble to clinicians and patients. Moreover, the value of conventional ultrasound in the differential diagnosis of breast masses is still limited, while the emergence of new technologies such as artificial intelligence and elastic imaging has improved the accuracy of ultrasound diagnosis to varying degrees.

The recently developed ultrasound light scattering imaging technology is used in breast ultrasound imaging systems to assist in morphological analysis based on the description and final evaluation of the Breast Imaging Reporting and Data System (BI-RADS), providing a new way to distinguish benign and malignant breast nodules.

Ultrasonic light scattering imaging technology is a new functional imaging technology that integrates traditional B-type ultrasound imaging and light scattering tomography (DOT). It uses B-type ultrasound to locate lesions and uses DOT to measure the concentrations of total hemoglobin, oxygenated hemoglobin and deoxygenated hemoglobin in diseased tissues based on the differences in the absorption rates of light of specific wavelengths in different tissues. It also measures the neovascularization at the tumor site and its potential local hypoxia stimulation. It introduces additional physiological information to current breast screening methods, often before morphological abnormalities. It can improve the accuracy of early diagnosis of breast cancer based on the characteristics of abnormal blood supply and oxygen consumption in lesions.

ELIGIBILITY:
Inclusion Criteria:

Had breast lesions detected by ultrasound Age 18 or older Upcoming FNAB or surgery Signing informed consent

Exclusion Criteria:

Patients who had received a biopsy of breast lesion before the ultrasound examination Can not cooperate with the test operation Patients who were pregnant or lactating Patients who were undergoing neoadjuvant treatment.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: In order to verify that ultrasound light scattering imaging technology can help in the differential diagnosis of benign and malignant breast nodules. For subjects who meet the inclusion criteria, breast nodules will be examined by traditional ultrasound and ultrasonic light scattering imaging, and the diagnostic efficacy of both will be determined based on the final pathological results of the subjects.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Benign breast tumor | Up to 12 months
  Pathological diagnosis
Malignant breast tumor | Up to 12 months
  Pathological diagnosis
Breast lymph node metastasis | Up to 12 months
  Pathological diagnosis
No lymph node metastasis | Up to 12 months
  Pathological diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Xin-Wu Cui, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang Y, Cua M, Brake J, Liu Y, Yang C. Investigating ultrasound-light interaction in scattering media. J Biomed Opt. 2020 Feb;25(2):1-12. doi: 10.1117/1.JBO.25.2.025002. PMID 32103649
- [Background] Di Sciacca G, Maffeis G, Farina A, Dalla Mora A, Pifferi A, Taroni P, Arridge S. Evaluation of a pipeline for simulation, reconstruction, and classification in ultrasound-aided diffuse optical tomography of breast tumors. J Biomed Opt. 2022 Mar;27(3):036003. doi: 10.1117/1.JBO.27.3.036003. PMID 35332743
- [Background] Zhu Q, Ricci A Jr, Hegde P, Kane M, Cronin E, Merkulov A, Xu Y, Tavakoli B, Tannenbaum S. Assessment of Functional Differences in Malignant and Benign Breast Lesions and Improvement of Diagnostic Accuracy by Using US-guided Diffuse Optical Tomography in Conjunction with Conventional US. Radiology. 2016 Aug;280(2):387-97. doi: 10.1148/radiol.2016151097. Epub 2016 Mar 2. PMID 26937708